CLINICAL TRIAL: NCT02865512
Title: An Analysis of Thoracic Epidurography Contrast Patterns According to Two Different Position of Patient
Brief Title: Thoracic Epidurography Different Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Associate professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-05-036
Record Dates: First submitted 2016-08-04; First posted 2016-08-12 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Thoracic Epidural Injection
Keywords: thoracic epidural injection; patient position

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- supine position (Active Comparator): thoracic epidural catheterization with supine position
  Interventions: Procedure: thoracic epidural catheterization
- flexed lateral position (Active Comparator): thoracic epidural catheterization with flexed lateral position
  Interventions: Procedure: thoracic epidural catheterization

INTERVENTIONS:
Procedure: thoracic epidural catheterization — thoracic epidural catheterization for the management of postoperative pain

SUMMARY:
It is known that postoperative pain after thoracotomy or lobectomy is very severe, therefore, intraoperative or postoperative pain management using continuous thoracic epidural catheterization is suggested good option to prevent this complication.

The spread of local anesthetics is influenced by various factors including volume, location of needle insertion, speed of injection, patient position, age, weight and height. However, there are few studies about the effect of different patient position during thoracic epidural catheterization.

This study was designed to evaluate the effect of different patient position affecting thoracic epidurography.

DETAILED DESCRIPTION:
It is known that postoperative pain after thoracotomy or lobectomy is very severe, therefore, intraoperative or postoperative pain management using continuous thoracic epidural catheterization is suggested good option to prevent this complication.

The spread of local anesthetics is influenced by various factors including volume, location of needle insertion, speed of injection, patient position, age, weight and height. However, there are few studies about the effect of different patient position during thoracic epidural catheterization.

Studies of lumbar epidural blockade have shown that lateral position can produce 0-3 segment more to the dependent position compared to the supine position. When the same amount of local anesthetic was injected in supine of sitting position, the most cephalad level of spread was indifferent.

Recent studies showed that neck flexion demonstrated significant cephalad spread of contrast dye in high thoracic epidural blockade.

The purpose of this study was to compare and evaluate the contrast dye spread between different patient position

ELIGIBILITY:
Inclusion Criteria:

* lung cancer
* liver cancer
* stomach cancer
* pancreas cancer

Exclusion Criteria:

* coagulopathy
* infection
* previous spine fusion at thoracic level

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Number of segment convered by contrast dye assessed through fluoroscopic image | 1 minutes after the completion of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hee Hong, MD, PhD, Principal Investigator — Keimyung University Dongsan Medical Center
Locations (1):
- Ji Hee Hong, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hong JH, Jung SW, Park JH. Posture Influences the Extent of Spread of Contrast Medium During Thoracic Epidurography: A Prospective Randomized Trial. Pain Physician. 2017 Sep;20(6):501-508. PMID 28934781